CLINICAL TRIAL: NCT05311917
Title: To Compare Home Vision Therapy and Prism Prescription in Presbyopic Persons With Convergence Insufficiency
Brief Title: Home Vision Therapy and Prism Prescription in Presbyopic Persons With Convergence Insufficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saeid Abdi, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1400.610
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Convergence Insufficiency
Keywords: vision therapy; prism prescription; convergence insufficiency
MeSH Terms: conditions — Ocular Motility Disorders | interventions — Alkalies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- home vision therapy (Experimental): near glasses will be prescribed along with a complete training of the exercises and with a eye exercise form of information about how and how long to do the exercise, by optometrist No 2 (Saeid Abdi).training includes: Voluntary convergence, Bug on string, Eccentric Circles, Jumping vergence , Barrel card, chiastopic fusion, Brock string, push-up These exercises will be done 3 days a week for 20 minutes ( 10 minutes at noon and 10 minutes at night ) for 2 month. Home exercises include eight vision therapy exercises and patients will do two exercises each day at noon and two exercises at night.
  Interventions: Other: home vision therapy
- base in prism prescription (Experimental): base in prism prescription using sheards criterion near prismatic glasses will be prescribed and the amount of prism will be divided between two eyes; and random and aimless eye movements, without convergence and accommodation effects will be prescribed by optometrist No. 2 (Saeid Abdi). patients should complete their checking form for eye exercises.
  Interventions: Other: base in prism prescription
- conventional (Placebo Comparator): new near glasses as a conventional treatment with the practice of random and aimless eye movements, without convergence and accommodation effects will be prescribed by optometrist No. 2 (Saeid Abdi). patients should complete the form of their eye training.
  Interventions: Other: conventional placebo

INTERVENTIONS:
Other: home vision therapy — a group of vision therapy procedures in home to improve convergence insufficiency
  Other Names: home eye training
  Arms: home vision therapy
Other: base in prism prescription — base in prism prescription according to sheards criterion
  Other Names: prism prescription
  Arms: base in prism prescription
Other: conventional placebo — using near glasses with aimless eye training
  Other Names: placebo
  Arms: conventional

SUMMARY:
convergence insufficiency is one of the most common binocular vision problems in which the eyes tend to have more exophoria in near than distance activities. Its prevalence is typically reported from 2.25% to 29.6% depending on the study population and its definition. Most of its symptoms include difficulty seeing at close works, headache, eye pain during study, blurred vision, diplopia, movement of words in reading, a feeling of pressure in the eye, and lack of concentration. Its signs include increasing near point of convergence, more exophoria at near than distance, decreased AC / A ratio, decreased positive fusional vergence.

In patients with convergent insufficiency, the first valid and standard questionnaire to assess the frequency and type of symptoms used before and after convergence insufficiency treatment is the convergence insufficiency symptom survey (CISS) questionnaire.

Generally, vision therapy is the first choice for convergence insufficiency management and the other choice is base in prism prescription. On the other hand, due to the changes in the interaction of the accommodation and convergence systems with increasing age, It is necessary to study how these systems interact and compare their responses to the active treatment of vision therapy and inactive prescription of base in prism.

In this controlled study, investigators will evaluate and compare the effect of vision therapy and base in prism prescription in patients over 40 years of age. this investigation will help to clarify which treatment is more effective.

This study will have two phases. In the first phase, investigators will seek to check the reliability and validity of the Persian version of CISS questionnaire for the elderly patients. For this purpose, investigators will use the Persian version questionnaire in previous study that assessed for young adults, and the investigators will modify it and check the reliability and validity of the final Persian version for subjects with presbyopia. This modified CISS questionnaire will be investigated in the elderly participants and the appropriate cut off point to differentiate between the normal group and the group with convergence insufficiency will be determined.

in the second phase one optometrist (Z.K.R) will do the preliminary examination and another optometrist (S.A) will do the interventions. After the initial examination and having the inclusion criteria, patients will be invited to participate in the study, the nature of the research will be explained to subjects and informed consent will be obtained from them. Before randomization, patients are asked to complete the CISS questionnaire and submit this questionnaire to Optometrist No. 1 (Z.K.R).According to the randomization all patients will be assigned to one of the treatment or control groups by optometrist No. 1. Vision therapy exercises, necessary trainings and prescriptions are given to all patients by Optometrist No. 2 (S.A).For the participants in the control group only near glasses will be prescribed as a conventional treatment, for the second group near glasses with base in prism according to sheard's criterion will be prescribed and in the third group, the prescription of near glasses will be given along with the complete training of the home exercises.

DETAILED DESCRIPTION:
Between non-strabismic binocular vision problems, convergence insufficiency is the most common problem (6) even in people with presbyopia this problem has high prevalence. (11) The most common ocular finding in these patients is an increase in near exophoria and thus reduces person's performance in activities such as reading, computer working and near activities. (12) Despite the effectiveness of vision therapy in reducing patients' symptoms and improving visual function, the different accommodation and vergence systems in the elderly may cause different results (1) so a comprehensive study of adult patients over the age of 40 with convergence insufficiency is needed. According to our knowledge the only study in these patients was done by MH Birnbaum (13) in 1999 which had several limitations. For example, in their study, the results were classified and recorded as success and failure in functional therapy and improvement or non-improvement of asthenopia; Success in treatment was achieved when two criteria were met: 1. The criterion of asthenopia includes achieving the ability to study for at least one hour without diplopia; And the ability to study without headache, eye pain and loss of concentration at least 75% of the time 2- Achieving 3 options of functional criteria including having an appropriate near point of convergence, having appropriate near point of convergence with red lens, having low near phoria and positive fusional vergence.

Another problem of this study was: not using the CISS questionnaire, which is a valid questionnaire of convergence insufficiency, and only considered success in treatment based on the two criteria, it should be mentioned that in their study the method for patients' selection did not report; On the other hand, the study was not blind, the importance of designing blind studies has been proven. Only one study by B Teitelbaum assessed prism prescription in patients over 40 years with convergence insufficiency (14) their study had two main problems, first: selected patients did not necessarily have convergence insufficiency, because the two basic criteria for convergence insufficiency (near point of convergence and positive fusion vergence) did not include in their study. Second: not using commercial progressive add lenses in patients glasses and it was unique lens with special design with limitation in base in prism prescription.

Because of the effects of various factors on vision therapy including patients' motivation, lack of cooperation in eye exercise, inappropriate age and unfavorable economic conditions, (especially in developing countries like Iran) or pandemic condition like COVID19 pandemy, vision therapy may not always be possible (1-3) and clinicians may have to prescribe base in prism for these patients. On the other hand, due to the changes in accommodation and convergence system and their interaction with aging (1, 3-4) study of their responses to the two types of treatments including active vision therapy and passive base in prism therapy and comparing them are noticeable matter and solving this challenge is absolutely necessary.

This study includes two phases. In the first phase, investigators will evaluate the reliability and validity of the Persian version of questionnaire for the elderly patients, this version was validated for young patients (38). Investigators will modify this questioner for presbyopic patients. For this purpose, six optometrists experienced in binocular vision will assess the questioner in two aspects: validity and reliability.

The validity of the modified Persian CISS include face validity (use of meaningful words), content validity (relevancy, clarity, comprehensiveness), discriminant validity Using a 6-point Likert scale (very weak, weak, moderate, good, very good, best), face validity will be assessed according to the aspects of fluency in elderly patients' cultural acceptance in iran and a score of ≥4 for each question will be passable. Content validity will be determined based on 1-relevancy (the extent to which the question of interest can being closely connected or appropriate for characteristics of the content under study), 2-clarity (appropriateness of the selected items in terms of being coherent and intelligible in concept and writing style), and 3-comprehensiveness (the ability of the questioner to cover all domains related to the topic under study). Relevancy and clarity will be assessed item by item and for the whole items in the questioners using a 4-point Likert scale (1-undesirable, 2-relatively desirable, 3-desirable, 4-completely desirable), and the Item Content Validity Index (I-CVI) and Scale Content Validity Index (S-CVI) will be calculated for the indices. Universal agreement approach will be used to check, the I-CVI value and it will be between 0-100%, and I-CVI≥ 0.8 will be considered passable. 20 The S-CVI for relevancy and clarity will be determined by averaging all I-CVI values. Comprehensiveness will be only measured at the scale level using a 4-point Likert scale (1- incomprehensive, 2- relatively comprehensive, 3- comprehensive, and 4- totally comprehensive). Then, the reliability of the questionnaire will be assessed using test-retest reliability analysis between first and second questioner administration in a group of 50 presbyopic patients aged 40-60 with convergence insufficiency. The elderly participants will be asked to participate in a second administration of the questionnaire 7-14 days later. To assess discriminant validity, convergence insufficiency will be categorized to 3 groups of mild (PFV ≥1.50 × near exophoria), severe (PFV < near exophoria), and moderate (values in between these groups) based on the severity of clinical manifestations according to the Convergence Insufficiency Treatment Trial guideline, and the mean overall CISS score Will be compared between these three groups.

Also, to evaluate the validity and reliability of the CISS questionnaire in the elderly patients and to determine the appropriate cut off point to differentiate between the normal group and the group with the problem of convergence insufficiency, a group of 50 people aged 40-60 with normal binocular vision to compare the scores will be considered to fill out the questionnaire and participants will complete the questionnaire again within 7 to 14 days.

T-test will be used to compare the scores of the convergence insufficiency group and the group with normal binocular vision; The area under the ROC curve will also be used to assess the ability of CISS scores to differentiate between individuals with convergence insufficiency and individuals with normal binocular vision. Intraclass Correlation Coefficient (ICC) will be used to assess the reliability of the CISS questionnaire.

In the second phase, After the initial examination and having the inclusion criteria, patients will be invited to participate in the study, all the steps and nature of the research will be explained to them and informed consent will be obtained from them. We will have two optometrists, all patients will be assigned to one of the treatment or control groups by optometrist number (1) (Zahra Kamary Rad). Before randomization, patients will be asked to complete the CISS questionnaire and submit this questionnaire to Optometrist No.1. Optometric examinations will be done by optometrist No1 (Zahra Kamary Rad) . First distance and near uncorrected visual acuity will be measured, then patients refraction will be measured by autokeratorefractometer (TOPCON, KR8800, Japan) and refraction will be repeated by retinoscope(beta 200 Heine Germany ). Subjective refraction with positive maximal lens method with maximum visual acuity will be obtained, distance heterophoria will be measured at six meters with covzer and prism bar and target two lines above the best visual acuity. The best visual acuity will be measured with near glasses at a distance of 40 cm and the cover test results are repeated three times and bracketing method will be used to determine the final result of the heterophoria measurements. The near point of convergence will be evaluated by red-green filters method. In this method the near point of convergence will be measured three times and the results will be averaged. The near point of convergence is recorded based on break and recovery point with near glasses. The amplitude of monocular accommodation will be calculated by push-up method, first in the right eye and then in the left eye.

Near step PFV will be measured by base out prism bar using 20/30 column at 40 cm with patients near glasses. Near vergence facility will be evaluated by flipper prism (3 base in and 12 base out) with target two lines above the best near-corrected visual acuity. This test will be also recorded by the patient's near glasses.

Stereopsis will be evaluated by the patients near glasses and red-green filters using TNO test. To check the prism adaptation, one hour after wearing the glasses, the amount of heterophoria will be measured again and the amount of change in the heterophoria is recorded as prism adaptation in percentag. Tropicamide 1% will be then dropped twice 5 minutes apart, in both eyes, and twenty minutes after the second drop refraction will be repeated; An ophthalmologist will check and confirm the health status of the eyes with a slit lamp and a +90 lens. After examining the patients by optometrist No. 1 vision therapy exercises and necessary trainings will be given to all patients by optometrist No. 2 (Saeid Abdi) In order to assign patients to each of the randomized treatment groups based on blocks classified according to age, gender and severity of convergence insufficiency.

For patients in control group new near glasses as a conventional treatment with the practice of random and aimless eye movements, without convergence and accommodation effects will be prescribed by optometrist No. 2 (Saeid Abdi) in Patients with base in prism prescription using sheards criterion near prismatic glasses will be prescribed and the amount of prism will be divided between two eyes; and random and aimless eye movements, without convergence and accommodation effects will be prescribed by optometrist No. 2 (Saeid Abdi).

In patients in the home exercise group , near glasses will be prescribed along with a complete training of the exercises and with a form of information about how and how long to do the exercise, along with random and aimless eye movements, by optometrist No 2 (Saeid Abdi).

These accommodation/ convergence training includes:

Voluntary convergence, Bug on string, Eccentric Circles, Jumping vergence , Barrel card, chiastopic fusion, Brock string, push-up These exercises will be performed by the patient in a variety of ways in each session. Which will be 3 days a week for 20 minutes ( 10 minutes at noon and 10 minutes at night ) and must record these exercises for 2 month. Home exercises include eight vision therapy exercises and patients willdo two exercises each day at noon and two exercises at night. Also, each exercise will be done five minutes , so subjects have to do four different exercises every day, and in the next session participants have to do the next four exercises.

Participants should register these trainings in a special form for 2 months. The total number of training sessions will be two months( 24 sessions) All prescribed glasses will be checked and used after confirmation, and patients do not know in which group categorized.

Practice and use of glasses will continue for 2 months and the participants will refer for the final examination and all optometric examinations will be repeated by optometrist No. 1 It should also be noted that base in prism will be prescribed according to the sheards criterion and will be rounded upwards and this amount of prism is evenly divided between the two eye.

ELIGIBILITY:
Inclusion Criteria:

CISS score more than the estimated cut off point

Best corrected visual acuity=20/20 for near and far

Having Convergence Insufficiency

Near exophoria should be at least 4 prisms more than distant exophoria

NPC more than 6 cm

Inadequate near-positive positive fusion according to the Convergence Insufficiency Treatment Trial (CITT) study (8)

Normal monocular accomodation amplitude according to Hofster formula

Exclusion Criteria:

Any type of strabismus

Amblyopia

Refractive error more than 6 diopters

Patients with history of prism prescription

History of vision therapy from 5 years ago

History of strabismus surgery or refractive error surgery

History of eye trauma

Use of any ophthalmic or general ophthalmic drugs affect ocular accommodation such as phenylephrine, anticholinergic drugs (mydriatics), carbonic anhydrase inhibitors, antihistamines, morphine and its derivatives, antidepressants amphetamine and imipramine

More than one prism of vertical phoria

Any mechanical limitations in the eye muscles

Ocular muscle paralysis

Nystagmus

Any systemic and neurological diseases affecting binocular vision such as diabetes, myasthenia gravis, Graves', multiple sclerosis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-04-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
treatment success criteria | 2 month after intervention
  achieving near point of convergence below 6 cm or 4 cm reduction in its distance, positive fusional vergence according to sheard criterion or grater than 15 prism or 10 prism improvement.
  achieving normal limit in CISS or 10 score improvement in total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti University of Medical Sciences, Tehran, Iran

REFERENCES:
- [Derived] Abdi S, Kangari H, Rahmani S, Baghban AA, Rad ZK. Home vision therapy and prism prescription in presbyopic persons with convergence insufficiency: study protocol for a randomized controlled trial. BMC Ophthalmol. 2024 Apr 15;24(1):169. doi: 10.1186/s12886-024-03411-y. PMID 38622543